CLINICAL TRIAL: NCT06506799
Title: "Determining the Effect of the Training Given to Intensive Care Nurses on Their Knowledge Level, Attitudes and Practices Regarding the Use of Physical Restraints"
Brief Title: Effect of Training on the Use of Physical Restraints
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Ogr. Uyesi Naile, Assistant Professor, Fenerbahce University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 66.2024fbu
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Fixation Device; Complications; Nursing Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Other): Data will be collected with the 'Participant Information Form' and the 'Nurses' Knowledge Level, Attitudes and Practices Regarding Physical Restraint Scale', prepared by the researcher in line with the literature and containing the demographic characteristics of the participants.
  Intensive care nurses who will participate in the research will be asked to fill out the survey forms with individual consent.
  Participant Information Form and Nurses' Knowledge, Attitude and Practice Levels Regarding Physical Restraint Scale will be used as pre-tests. After the pre-test, nurses will be given physical restraint training. The training content was created using the ADDIE model as reference. After the training, the Nurses' Knowledge Level, Attitudes and Practices Regarding Physical Restraint Scale will be used as the final test.
  Interventions: Other: Training Given to Intensive Care Nurses on the Use of Physical Fixation

INTERVENTIONS:
Other: Training Given to Intensive Care Nurses on the Use of Physical Fixation — Data will be collected with the 'Participant Information Form' and the 'Nurses' Knowledge Level, Attitudes and Practices Regarding Physical Restraint Scale', prepared by the researcher in line with the literature and containing the demographic characteristics of the participants.
  Intensive care nurses who will participate in the research will be asked to fill out the survey forms with individual consent.
  Participant Information Form and Nurses' Knowledge, Attitude and Practice Levels Regarding Physical Restraint Scale will be used as pre-tests. After the pre-test, nurses will be given physical restraint training. The training content was created using the ADDIE model as reference. After the training, the Nurses' Knowledge Level, Attitudes and Practices Regarding Physical Restraint Scale will be used as the final test.

SUMMARY:
Patients in the intensive care unit may harm themselves by pulling medical equipment such as endotracheal tube, monitoring, arterial and peripheral catheters. Physical detection is also one of the common practices used in this case. Physical restraint is a practice performed by using patient aids to protect the individual or other patients around him, to ensure his safety and to control his behavior. Although physical detection seems to be a useful and simple method, it brings with it various physical, psychological, ethical, legal and moral problems. Nurses should use alternative strategies to prevent and reduce the use of restraint, and to avoid the negative consequences that may be caused by restraint by performing restraint appropriately and effectively, and thus ensure the safety of the patient. Evaluating nurses' knowledge on this subject, identifying deficiencies and providing training is important in terms of improving the quality of care and ensuring patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in an adult intensive care unit
* Fill out the form completely
* Volunteering to participate in the study
* No vision or language problems to fill out the form

Exclusion Criteria:

* Filling the form incompletely
* Coming to the intensive care unit on rotation
* Not attending training
* No vision or language problems to fill out the form
* Having previously received training on physical detection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-08-28 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
outcome 1 | 2 week
  Training on the Use of Physical Restraint Given to Intensive Care Nurses Will Increase the Score of the Nurses' Knowledge Level, Attitudes and Practices Regarding Physical Restraint Scale.

IPD SHARING:
Plan to Share IPD: No